CLINICAL TRIAL: NCT06962696
Title: Assessing the Performance of GPT-4o in Evaluating the Safety of Home Environment for Older Adults
Status: Recruiting | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M20241058
Record Dates: First submitted 2025-02-10; First posted 2025-05-08 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-01

CONDITIONS: Elderly (People Aged 65 or More); Home Environment Related Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: No intervention — no intervention provided

SUMMARY:
This study is an investigative study, taking the elderly in Beijing community as an example, and taking photos of different areas in the home environment of the elderly who agree to participate in the study (a total of seven aspects, including pathways/entrance to home, hallways, stairs/steps, living room, kitchen, restroom, bedroom). Subsequently, the multi-modal large model GPT-4o and a professional occupational therapist will use the "Home Environment Assessment" scale to evaluate the home environment shown in the photos and give corresponding suggestions for modification. A professional occupational therapist (non-evaluator) will analyze and compare the evaluation results and guidance recommendations of GPT-4o and the evaluator, and compare whether there are any significant differences between the two analysis results.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥65 years old
2. Staying in the place of residence for a long time
3. Having normal listening, speaking, and comprehension skills

Exclusion Criteria:

Does not live regularly in the place of residence

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: The elderly are older than or equal to 65 years old, regardless of gender, and have been living in Beijing for a long time.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Home Environment Assessment Scale | 1 day
  Use the "Home Environment Assessment" scale to evaluate the aging suitability of the home environment of enrolled older adults. The scale can assess a total of seven places, including pathways/entrance to home, hallways, stairs/steps, living room, kitchen, restroom, bedroom.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China